CLINICAL TRIAL: NCT04956978
Title: Shared Decision Making to Address Racial Disparities in Oral Anticoagulation Use in Patients With Non-valvular Atrial Fibrillation
Brief Title: Shared Decision Making to Address Racial Disparities in Oral Anticoagulation in NVAF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00108334
Record Dates: First submitted 2021-06-25; First posted 2021-07-09 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation
Keywords: Oral Anticoagulation; Health Disparities
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Decision Support Tool (Experimental): Patient decision support tool to be used in conjunction with physician counseling to discuss the risk and benefits of systemic oral anticoagulation.
  Interventions: Other: Patient Decision Support Tool
- Usual Healthcare Counseling (No Intervention): Traditional physician counseling regarding the risk and benefits of systemic oral anticoagulation

INTERVENTIONS:
Other: Patient Decision Support Tool — Patient decision support tool is a web based educational material that informs a patient on the risk and benefits of oral anticoagulation. In addition, such a tool aims to assess patient values and preferences in the decision making process for oral anticoagulation for stroke reduction.
  Arms: Patient Decision Support Tool

SUMMARY:
The study is a pilot analysis using a decision on the risk and benefits of oral anticoagulation for stroke reduction for patients with non-valvular atrial fibrillation. This study is a feasibility and acceptability analysis but will also measure preliminary effectiveness measures.

The investigator hypothesizes that a patient decision support tool will increase decision quality and secondarily increase the use of oral anticoagulation in Black patients with non-valvular atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Black and White adults greater than or equal to 18 years of age
* Clinical diagnosis of NVAF
* CHA2DS2-VASc score greater than or equal to 2
* New patient visit for initiation of oral anticoagulation at primary care and cardiology clinics

Exclusion Criteria:

* Unable to speak English
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients willing to consent as measured by enrollment log | End of Study, 12 months
Proportion of patients willing to participate as measured by enrollment log | End of Study, 12 months
Rate of completion of questionnaire measures as measured by Research Electronic Data Capture (REDCAP) | End of Study, 12 months
  Measured by RedCap (all questionnaires will be distributed through RedCap)
Rate of Patient Decision Support tool delivery and data capture as measured by web based data capture | End of Study, 12 months
Percent of patients who stated that the intervention was acceptable as measured by patient and provider interviews. | 1 week post clinic visit

SECONDARY OUTCOMES:
Decision Quality measured by use of the decision conflict scale | Clinical Day, up to 1 day
Decision to initiate systemic oral anticoagulation measured and documented by physician of record during clinic visit. | Clinical Day, up to 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Larry Jackson, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No